CLINICAL TRIAL: NCT03868319
Title: Effect of Lung-protective Ventilation During Robot-assisted Laparoscopic Radical Cystectomy on Postoperative Pulmonary Complication
Brief Title: Lung-protective Ventilation During Robot-assisted Laparoscopic Radical Cystectomy
Acronym: LPV-RARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, DAN HUANG, Principal Investigator, clinical attending in anesthesia department, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Da vinci
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Lung-protective Ventilation
Keywords: lung-protective ventilation strategy; low tidal volume; positive end-expiratory pressure; Lung ultrasound; postoperative pulmonary complications

STUDY DESIGN:
Intervention Model Description: Lung-protective ventilation(LPV) group (low tidal volume 6 ml kg-1 predicted ideal body weight (PBW)+ 7 cmH2O positive end-expiratory pressure(PEEP)) vs. nonprotective group (control group) (large tidal volume 9 ml kg-1 + zero PEEP (ZEEP)) mechanical ventilation in patients undergoing RARC
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators, surgeons and patients remained unware of study-group assignments so as to preserve the double blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): nonprotective ventilation with a tidal volume of 9 ml kg-1 PBW with ZEEP
  Interventions: Procedure: nonprotective ventilation
- LPV group (Experimental): a tidal volume of 6 ml kg-1 PBW with a 7 cmH2O level PEEP
  Interventions: Procedure: lung protective ventilation strategy

INTERVENTIONS:
Procedure: lung protective ventilation strategy — low tidal volumes and positive end-expiratory pressure mechanical ventilation during robot-assisted laparoscopic radical cystectomy for bladder cancer
  Arms: LPV group
Procedure: nonprotective ventilation — large tidal volume and zero PEEP mechanical ventilation during robot-assisted laparoscopic radical cystectomy for bladder cancer
  Arms: control group

SUMMARY:
Robot-assisted laparoscopic radical cystectomy (RARC) increases the incidence of postoperative complications. We conducted a study to determine the effect of lung-protective ventilation strategy.

DETAILED DESCRIPTION:
Robot-assisted laparoscopic radical cystectomy (RARC) performed with patient in the steep Trendelenburg position under pneumoperitoneum increases the incidence of postoperative complications. Approach termed lung-protective ventilation (LPV) strategy which refers to the use of low tidal volumes and positive end-expiratory pressure (PEEP) may lead to a reduction in inflammation and prevent the occurrence of atelectasis. Computed tomography (CT) requiring transportation is the golden standard for measuring atelectasis, which is not suitable for perioperative observation. Lung ultrasound (LUS) which is noninvasive and easily repeatable at the bedside appears to be an accurate diagnostic tool for early detection of atelectasis. Thus, we conducted the trial to determine whether an LPV strategy has benefits in patients scheduled for RARC through a multifaceted method. We hypothesized that the use of prophylactic low tidal volume and PEEP would decrease postoperative inflammation and atelectasis, thereby, improve outcomes, as compared with the standard of nonprotective mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective RARC

Exclusion Criteria:

* history of lung surgery
* patients' refusal or inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
occurrence of postoperative pulmonary complications (PPCs) | during the first 90 days after surgery
  graded on a scale from 0 (no pulmonary complications) to 4 (the most severe complications)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xie, PhD, Study Chair — The Second Affiliated Hospital of Soochow University, China
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China